CLINICAL TRIAL: NCT00672165
Title: Phase I Trial of Targeted Atomic Nano-Generators (Actinium-225-Labeled Humanized Anti-CD33 Monoclonal Antibody HuM195) in Patients With Advanced Myeloid Malignancies
Brief Title: Targeted Atomic Nano-Generators (Actinium-225-Labeled Humanized Anti-CD33 Monoclonal Antibody HuM195) in Patients With Advanced Myeloid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Actinium Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-017; NCI CA33049
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: MAB HUM 195 ACTINIUM-225 LABELED; HEMATOPOIETIC SYSTEM; 02-017
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes

ARMS (1):
- 1 (Experimental): This is a phase I, dose-escalation trial. The starting dose level will be 0.5 μCi/kg of 225Ac-HuM195. Three to six patients will be treated at each dose level, and dose escalation will proceed if less than 33% of patients in a cohort experience dose limiting toxicity. Six patients will be treated at the maximum tolerated dose
  Interventions: Biological: ACTINIUM-225-LABELED HUMANIZED ANTI-CD33 MONOCLONAL ANTIBODY HuM195

INTERVENTIONS:
Biological: ACTINIUM-225-LABELED HUMANIZED ANTI-CD33 MONOCLONAL ANTIBODY HuM195 — A single infusion of 225Ac-HuM195 will be administered at a starting dose of 0.5 μCi/kg. Additionally, 100 mCi of 213Bi-HuM195 have been administered with full dose cytarabine (200 mg/m2 daily for 5 days) without dose-limiting toxicity.Serial sampling of blood, urine, and bone marrow will be performed following treatment to determine the toxicity, pharmacokinetics, immunogenicity, and antileukemic effects. Three to six patients will be treated at each dose level. Dose escalation will proceed if less than 33% of patients in a cohort experience dose-limiting toxicity.Patients will be followed until completion of therapy as outlined in the study, loss to follow-up, death, or until the day the patient is removed from the study.

SUMMARY:
The purpose of this study is to find a safe dose of actinium-225 when it is labeled to HuM195. This will be done with a "phase I trial," in which a preset schedule of doses gets more powerful for each new group of patients as the trial progresses. If too many serious side effects are seen with a certain dose, no one will be treated with a higher dose, and some additional patients may be treated with a lower dose to make sure that this dose is safe. The starting dose of actinium-225 in this study is less than doses that are known to be safe in animals.

Antibodies are proteins that are produced by the immune system and help the body to fight foreign substances, such as bacteria or viruses. HuM195 was made by putting human leukemia cells into mice. Most of the mouse parts of this antibody were replaced with human parts. Only the part of the antibody that binds to the leukemia cells was kept from the mouse. HuM195 attaches to leukemia cells but does not attach to most normal cells. It can kill small amounts of disease by identifying the leukemia cells as "foreign." HuM195 has worked less well against large amounts of leukemia since the normal immune cells needed to kill leukemia cells are lowered in most patients with leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have one of the following pathologically confirmed diagnoses:
* AML in relapse,
* AML refractory to at least 2 courses of standard induction chemotherapy or one course of high-dose cytarabine-containing induction chemotherapy,
* CML in accelerated phase or myeloid blast crisis that has progressed after treatment with imatinib and a second generation tyrosine kinase inhibitor (e.g., dasatinib or nilotinib)
* RAEB with International Prognostic Scoring System (IPSS) score ≥ 2.5, or - CMMOL with IPSS score ≥ 2.5 refractory to or relapsed after a hypomethylating agent (e.g., azacitidine or decitabine) refractory to or relapsed after a hypomethylating agent (e.g., azacitidine or decitabine).
* Greater than 25% of bone marrow blasts must be CD33 positive.
* Patients must have a life expectancy of at least 6 weeks and a Karnofsky performance status of ≥ 60%.
* Adequate renal function as demonstrated by a serum creatinine ≤ 1.5 mg/dl, a creatinine clearance > 60 ml/min, and < 1 gram urinary protein/24 hours.
* Adequate hepatic function as demonstrated by a bilirubin ≤ 1.5 mg/dl (unless attributable to leukemia or Gilbert's disease) and alkaline phosphatase and AST ≤ 2.5 times the upper limit of normal.

Exclusion Criteria:

* Untreated AML, regardless of prognostic features.
* Treatment with chemotherapy or biologic therapy within 3 weeks of 225Ac- HuM195 administration. Hydroxyurea is permitted but must be discontinued prior to treatment on study. Patients must have recovered from the effects of previous treatment.
* Treatment with radiation therapy within 6 weeks of 225Ac-HuM195 administration. Patients must have recovered from the effects of previous treatment.
* Active serious infections not controlled by antibiotics.
* Pregnant women or women who are breast-feeding.
* Concurrent active malignancy requiring therapy.
* Clinically significant cardiac disease (NY Heart Association Class III or IV)or pulmonary disease.
* Patients with HLA-compatible donor bone marrow who are immediate candidates for bone marrow transplantation.
* Patients who are candidates for alternative treatments of known effectiveness.
* Patients eligible for protocols of higher priority.
* Patients previously treated with any monoclonal antibody for any reason.
* Active CNS leukemia
* Other serious or life-threatening conditions deemed unacceptable by the principal investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of 225Ac-HuM195 that can be administered to patients with advanced myeloid leukemias. | conclusion of study

SECONDARY OUTCOMES:
To determine the pharmacokinetics and dosimetry of 225Ac-HuM195. | conclusion of the study
To determine the biological effects of 225Ac-HuM195, including its ability to produce complete remissions. | conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Dan Douer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Nikitaki Z, Velalopoulou A, Zanni V, Tremi I, Havaki S, Kokkoris M, Gorgoulis VG, Koumenis C, Georgakilas AG. Key biological mechanisms involved in high-LET radiation therapies with a focus on DNA damage and repair. Expert Rev Mol Med. 2022 Mar 31;24:e15. doi: 10.1017/erm.2022.6. PMID 35357290
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org